### **Cover Page**

**Document Type:** Informed Consent Form

**Study Official Title:** The Effects of Stimulus Variability in Natural Visual Scenes

**Study NCT Number:** NCT05004649

**Document Date**: August 5, 2021

### UNIVERSITY OF PENNSYLVANIA

David Brainard, Department of Psychology (215) 573-7579

#### CONSENT FORM

Color Constancy and Visual Perception

**INVITATION TO PARTICIPATE**: You are being asked to participate in a research study on visual perception.

**PURPOSE**: The purpose of this experiment is to investigate how our visual system determines the properties of objects, and/or to explore more generally how light is processed by the human visual system.

**PROCEDURES**: You will look at a series of lights, objects, or images and make responses that indicate some aspect of what you see. You will make your response verbally, by pressing buttons, by manipulating a joystick, by typing at a keyboard, or in some similar fashion. In some experiments, your eye movements may be monitored and recorded. In some experiments you may be asked to fill in a series of brief questionnaires. The experimenter will give you specific information about what you will see and what you are expected to do.

**RISKS**: Participation in vision experiments of this kind involves no known risk to the subject. You may, however, become a bit bored or experience eye strain during the experimental session.

**COSTS AND FINANCIAL RISKS**: There are no known costs or financial risks associated with participation in this study.

**BENEFITS**: This study is part of a research program designed to advance our understanding of how vision works. There are no direct benefits to subjects participating in this study beyond the monetary compensation offered in return for participation.

**ALTERNATIVES**: Your participation in this study is completely voluntary. The alternative to participating in this study is not to participate in it. If at any point during the study you wish to terminate your participation, you are free to do so. You will be compensated for the time you actually spent participating in the study.

**PAYMENT**: You will be paid for your participation in this study at an hourly rate of \$15/hour. You will be paid for the time you actually participated, whether or not you complete the full study. In some studies, there may be a bonus payment that depends on the degree to which your visual judgments are objectively correct. The experimenter will review any such bonus with you as part of the instructions for the study. The bonus will not exceed \$15/hour.

**CONFIDENTIALITY**: Every attempt will be made by the investigators to maintain personal information collected in this study strictly confidential, except as may be required by court order or by law or as relevant to the presentation and interpretation of the data reported in presentations and publications. Authorized representatives of the University of Pennsylvania Institutional Review

### **CONSENT FORM**

### Color Constancy

Board (IRB), a committee charged with protecting the rights and welfare of research subjects, may be provided access to medical or research records that identify you by name. Data from this study may be reported in scientific presentations open to the public and publications available to the public. You will not be identified in such presentations or publications by name; single subject data may be presented but will be identified only by code number so people cannot tell that you participated nor which data are from you. Data collected in this study may also be released to the general public via a fully open database that may be accessed using the Internet. In the data that we share with the general public, subjects will again only be identified by code number, so people who access the data cannot tell that you participated nor which data are from you. No identifying information will be shared with the general public or anyone who is not laboratory personnel. Additionally, the data and samples contained within research records from this study might be used for other, future research projects in addition to the current study. These future projects can focus on any topic, and might have goals unrelated to those of this study. If you withdraw from the study we will cease data collection. However, any data and research results already collected may be used in presentations/publications, shared with the general public, or with other investigators. Once data has been presented, published, shared with the general public or other investigators it cannot be destroyed, withdrawn or recalled. You must be willing to have data from you shared in this way in order to participate in this study. If you are not willing to allow data from you to be shared in this way, you cannot participate in this study.

**ADDITIONAL INFORMATION**: Any significant new findings developed during the course of the study that may relate to your willingness to continue their participation will be provided to you.

**DISCLAIMER/WITHDRAWAL**: Your participation in this study is completely voluntary and that you may withdraw at any time without prejudicing your standing within the University of Pennsylvania or any class you might be taking.

**INJURY/COMPLICATIONS**: In the event of any physical injury resulting from the research procedures, medical treatment will be provided without cost to you, but financial compensation is not otherwise available from the University of Pennsylvania.

**SUBJECT RIGHTS**: If you wish further information regarding your rights as a research subject, you may contact the Director of Regulatory Affairs at the University of Pennsylvania by telephoning (215) 898-2614.

If you have any questions pertaining to your participation in this research study, you may contact the principal investigator by calling the telephone number listed at the top of page one.

You have been given the opportunity to ask questions and have had them answered to your satisfaction.

**CONCLUSION**: You have read and understand the consent form. You agree to participate in this research study. Upon signing below, you will receive a copy of the consent form.

## **CONSENT FORM**

# Color Constancy

| Name of Subject | Signature of Subject | Date/Time |
|---|---|---|
| Name of Person Obtaining<br>Consent | Signature of Person Obtaining Consent | Date/Time |